CLINICAL TRIAL: NCT04390477
Title: The Intestinal Microbiota as a Therapeutic Target in Hospitalized Patients With COVID-19 Infection
Brief Title: Study to Evaluate the Effect of a Probiotic in COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bioithas SL (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COVID.PROB
Record Dates: First submitted 2020-05-07; First posted 2020-05-15 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2021-07

CONDITIONS: COVID-19; Coronavirus Infection
Keywords: Probiotic
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — Probiotics

STUDY DESIGN:
Masking Description: Random numbers table. One branch placebo and other one no intervention
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Experimental): 1 pill od containing 1x10E9 cfu of the probiotic
  Interventions: Dietary Supplement: Probiotic
- Control (No Intervention): No treatment

INTERVENTIONS:
Dietary Supplement: Probiotic — Oral daily capsule containing probiotic strains with maltodextrin as excipient, administrated for 30 days.
  Arms: Probiotic

SUMMARY:
A prospective case-control pilot study to evaluate the possible effect of a probiotic mixture in the improvement of symptoms, the reduction in the number of days of hospitalization and the increase in the percentage of patients with negative PCR after infection with the coronavirus SARS-CoV-2.

DETAILED DESCRIPTION:
In this study, the investigators hypothesize a positive effect of probiotic on the gut microbiome that could led to produce a less severe clinical evolution of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a confirmed diagnosis of SARS-Cov.2 infection using the PCR and that require admission to the hospitalization area.

Exclusion Criteria:

* Inability or refusal to sign informed consent.
* Allergy or intolerance to the intervention product or its components.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2020-05-04 (Actual); Primary Completion 2021-03-21 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Cases with discharge to ICU. | 30-days
  Percentage of patients with discharge to ICU.
Patients with resolution of digestive symptoms | 30 days
  Percentage of patients with improvement between the initial and final visits

SECONDARY OUTCOMES:
Patients with home discharge. | 30-days
  Percentage of patients with home discharge.
Mortality. | 30-days
  Percentage of deaths.
Treatment safety assessed by number of adverse events. | 30-days
  Number of adverse events that occur during the treatment period, attributable or not to the intervention product.
New cases of SARS-Cov-2 infection among healthcare personnel caring for the patients. | 30-days
  Number of new cases of positive SARS-Cov-2 infection by PCR analysis.
Patients with negative PCR and/or Antigen test result for SARS-CoV-2 infection. | 10-15 days
  Percentage of patients with negative test for SARS-CoV-2.
Patients with resolution of non-digestive symptoms | 30 days
  Percentage of patients with improvement between the initial and final visits

CONTACTS AND LOCATIONS:
Overall Officials: Vicente Navarro, Principal Investigator — Hospital universitario del Vinalopo, Elche, Spain
Locations (2):
- Spain (2):
  - Hospital Universitario del Vinalopó, Elche, Alicante
  - Hospital Universitario de Torrevieja, Torrevieja, Alicante